CLINICAL TRIAL: NCT03836118
Title: Retrospective Evaluation of Clinical Predictors of Pregnancy and Live-birth After Homologous Intrauterine Insemination
Brief Title: Intrauterine Insemination Predictor Factors
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 7/18
Record Dates: First submitted 2019-02-08; First posted 2019-02-11 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IUI: all the IUI with controlled ovarian stimulation cycles in an academic tertiary ART center between January 1997 and December 2017
  Interventions: Procedure: Homologous intrauterine insemination (IUI)

INTERVENTIONS:
Procedure: Homologous intrauterine insemination (IUI) — Patients were treated with HMG/rFSH according to classic protocols of therapy and monitoring. An injection of uHCG 5000 IU/ rHCG 250 mg was given to trigger ovulation. On the day of insemination, the semen sample was obtained through masturbation after a 2-5 day abstinence period and collected in a sterile cup. TMSC was determined by multiplying grade A or grade A + B sperm motility percentages by sperm volume and concentration. To evaluate sperm viability Eosin and Nigrosin (E&N) staining was carried out according to WHO standards. Sperm capacitation was performed using density gradient centrifugation or swim-up procedure in order to remove seminal fluids and enhance sperm quality for IUI.
  IUI was performed a t36 hours post-HCG. A fraction of the washed motile spermatozoa was inserted up to the uterine fundus and expelled into the uterine cavity. Daily treatment with micronized progesterone was prescribed for 14 days after IUI. Serum ß-HCG was determined 14 days after IUI.

SUMMARY:
Multiple studies have reported on the impact of factors such as female age, duration of infertility, type of infertility, hormone levels (i.e. AMH, FSH, estradiol, progesterone), use of different ovarian stimulation protocols, timing/induction of ovulation, number of pre-ovulatory follicles, endometrial thickness by the time of ovulation, sperm parameters (i.e. concentration, progressive motility, morphology, total motile sperm count [TMSC], inseminating motile count [IMC]) and sperm washing procedures. Also the influence of body mass index and smoking on IUI outcome have been studied before. However, results on the predictive value of these parameters remain highly contradictory. The aim of the study is to examine the value of different variables in the prediction of IUI success to develop a clinically useful predictive model of pregnancy and live birth.

ELIGIBILITY:
Inclusion Criteria:

* couples had been diagnosed with infertility according to WHO definition (failure to achieve a clinical pregnancy after 12 months or more of regular unprotected sexual intercourse)
* at least one permeable tube
* a motile sperm concentration post treatment of 1×106/mL on the day of the semen analysis

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The included couples were subjected to an infertility diagnostic work-up. The tests included collecting medical history, physical examination, transvaginal ultrasound, serum hormone assays between day 2 and 4 of the menstrual cycle, semen analysis, uterine cavity and tubal patency evaluation with hysterosalpingography (HSG) or hysterosonosalpingography (HSSG) and/or hysteroscopy and video laparoscopy. Assessment of vaginal infection with cervico-vaginal swab and cultures
Sampling Method: Non-Probability Sample
Enrollment: 2970 (Actual)
Dates: Start 1997-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate (CPR) | 1997-2017
live-birth rate (LBR) | 1997 - 2017

CONTACTS AND LOCATIONS:
Locations (1):
- Paolo Emanuele Levi Setti, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Immediata V, Patrizio P, Parisen Toldin MR, Morenghi E, Ronchetti C, Cirillo F, Baggiani A, Albani E, Levi-Setti PE. Twenty-one year experience with intrauterine inseminations after controlled ovarian stimulation with gonadotropins: maternal age is the only prognostic factor for success. J Assist Reprod Genet. 2020 May;37(5):1195-1201. doi: 10.1007/s10815-020-01752-3. Epub 2020 Mar 25. PMID 32215826